CLINICAL TRIAL: NCT05402111
Title: A Randomized, Open-Label, Single Dose, Cross-over Study of Gastric Emptying Rate: SEP-363856 vs Prior Antipsychotic Standard of Care in Subjects With Schizophrenia
Brief Title: A Clinical Study That Will Assess How Food Moves Through the Stomach and Effects Blood Glucose Levels in Subjects With Schizophrenia Taking SEP-363856 or and Prior Antipsychotic (PA) Standard
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SEP361-124
Record Dates: First submitted 2022-05-24; First posted 2022-06-02 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856; Risperidone; Olanzapine; Quetiapine Fumarate; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SEP-363856 (Experimental)
  Interventions: Drug: SEP-363856
- Prior antipsychotic (risperidone, olanzapine, quetiapine or aripiprazole) (Active Comparator)
  Interventions: Drug: Prior antipsychotic (risperidone, olanzapine, quetiapine or aripiprazole)

INTERVENTIONS:
Drug: SEP-363856 — SEP-363856 will be supplied by 25 mg and 50 mg tablets. Multiple tablets may be required to achieve a single dose.
  Arms: SEP-363856
Drug: Prior antipsychotic (risperidone, olanzapine, quetiapine or aripiprazole) — PA will be prepared by the pharmacy staff according to the patient's prescribed treatment and will be orally administered. Multiple tablets or capsules may be required to achieve a single dose.
  Arms: Prior antipsychotic (risperidone, olanzapine, quetiapine or aripiprazole)

SUMMARY:
A clinical study to determine whether an investigational medication (SEP363856) changes how long it takes for food to move through the stomach into the small intestine in patients with schizophrenia. This study is accepting both male and female subjects. It will be conducted in approximately 6 study sites in the United States. The duration of participation will be approximtely 10 weeks.

DETAILED DESCRIPTION:
This is a randomized, open-label, single dose two-period crossover study with two treatment sequences. For each treatment sequence, subjects will receive a single-dose of SEP-363856 and prior antipsychotic (PA) standard of care (PA) in random order. Up to 3 separate cohorts of subjects will be randomized to determine the final dose of SEP-363856.

ELIGIBILITY:
Inclusion Criteria: (this list is not all inclusive)

* Male or female subjects between 18 and 65 years of age, inclusive at time of consent.
* Subject meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for a primary diagnosis of schizophrenia as established by clinical interview, using the DSM-5 as a reference and confirmed using the Structured Clinical Interview for DSM-5, Clinical Trials Version [SCID-CT]).
* Subject must have a CGI-S score ≤ 4 (normal to moderately ill) at Screening
* Subject must have a PANSS total score ≤ 80 at Screening and a score of ≤ 4 on the following PANSS items at Screening: P7 (hostility) and G8 (uncooperativeness)
* Subjects' antipsychotic medication at screening must have had no dose change (minor dose adjustments for tolerability purposes are permitted) for at least eight weeks prior to the Screening visit.

Exclusion Criteria: (this list is not all inclusive)

* Subject has a DSM-5 diagnosis or presence of symptoms consistent with a DSM-5 diagnosis other than schizophrenia or intellectual disability (IQ < 70).

  * Subject has attempted suicide within 12 months prior to Screening.
  * Subject answers "yes" to "Suicidal Ideation" Items 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS at Screening (ie. in the past 1 month) or at any subsequent C-SSRS assessment prior to dosing (ie, since last visit).
  * Subject is at risk of harming him/herself or others according to the Investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Gastric emptying T 1/2 (gastric emptying scintigraphy (GES) imaging) | multiple time-points post-radiolabelled meal on dosing day 1 and 2
  Gastric emptying T 1/2 (gastric emptying scintigraphy (GES) imaging) is gastric emptying half life (T1/2), which is a time needed for the half of the ingested gastric solids to leave the stomach.
Gastric retention at 4 hr post-radiolabeled meal (gastric emptying scintigraphy (GES) imaging) | 4 hours post-radiolabel meal on dosing Day 1 and 2
  Gastric retention at 4 hr post-radiolabeled meal is gastric retention 4h post meal, which estimates a percentage of remaining gastric solids in the stomach 4 hours after the meal.

SECONDARY OUTCOMES:
Gastric retention (proportion retained or % retained) at 1 hr and 2 hr post-radiolabeled meal | 1 and 2 hours post-radiolabel meal
  Gastric retention (proportion retained or % retained) at 1h and 2h post meal.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - CNRI - San Diego, LLC, San Diego, California
  - Galiz Research, Hialeah, Florida
  - Research Centers of America, Oakland Park, Florida
  - Pillar Clinical Research LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinical-trials.otsuka.com